CLINICAL TRIAL: NCT01674270
Title: Phase II Randomized Open Label Study of Neo-Adjuvant Degarelix vs. LHRH Agonist in Prostate Cancer Patients Prior to Radical Prostatectomy
Brief Title: Degarelix Neo-Adjuvant Radical Prostatectomy Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEG_PRE-OP_001; Degarelix Pre-Op
Record Dates: First submitted 2012-08-23; First posted 2012-08-28 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; bicalutamide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Degarelix (Experimental): Degarelix Alone
  Interventions: Drug: Degarelix
- Degarelix + Casodex (Experimental): Degarelix and Casodex
  Interventions: Drug: Degarelix; Drug: Casodex
- LHRH Agonist + Casodex (Active Comparator): LHRH Agonist and Casodex
  Interventions: Drug: Casodex; Drug: LHRH Agonist

INTERVENTIONS:
Drug: Degarelix
  Arms: Degarelix; Degarelix + Casodex
Drug: Casodex
  Arms: Degarelix + Casodex; LHRH Agonist + Casodex
Drug: LHRH Agonist
  Arms: LHRH Agonist + Casodex

SUMMARY:
To assess the effect of neo-adjuvant GnRH antagonist, degarelix, versus LHRH agonist on intratumoral levels of androgens.

ELIGIBILITY:
Inclusion Criteria:

* Men >18 and =< 75 years of age
* Willing and able to provide informed consent, either alone or with the aid of a translator
* Histologically confirmed prostate cancer as determined by transrectal ultrasound (TRUS) guided prostate biopsy performed within 6 months of study enrolment
* Gleason Score >= 7and/or prostate cancer that is clinical stage T2 disease.
* Candidates for open radical prostatectomy considered surgically resectable by urologic evaluation
* Normal organ and marrow function as defined by the following criteria:
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1

Exclusion Criteria:

* Previous or current use of hormonal management of prostate cancer (surgical castration or other hormonal manipulation, including GnRH receptor agonists, GnRH receptor antagonists, anti-androgens, estrogens, megestrol acetate, and ketoconazole)
* History of receiving radiation to the pelvic area.
* Previously received therapy with 5-alpha reductase inhibitors finasteride and/or dutasteride 4 weeks prior to randomization.
* History of bilateral orchiectomy, adrenalectomy, or hypophysectomy.
* History of severe untreated asthma, anaphylactic reactions, or severe urticaria and/or angioedema.
* Known hypersensitivity towards any component of the investigational medicinal product or Casodex (bicalutamide) or their excipients.
* Marked baseline prolongation of QT/QTcF interval (e.g. repeated demonstration of a QTcF interval >450 ms).
* History of risk factors for Torsade de Pointes ventricular arrhythmias (e.g. heart failure, hypokalemia, or family history of Long QT Syndrome).
* Previous history or presence of another malignancy, other than prostate cancer or treated squamous / basal cell carcinoma of the skin, within the last five years.
* Clinically significant laboratory abnormalities (e.g. severe renal or hepatic impairment) which in the judgment of the Investigator would affect the patient's health or the outcome of the trial.
* Clinically significant disorder (other than prostate cancer) including, but not limited to, renal, haematological, gastrointestinal, endocrine, cardiac, neurological, or psychiatric disease, and alcohol or drug abuse or any other condition, which may affect the patient's health or the outcome of the trial as judged by the Investigator.
* Use of natural medicines thought to have endocrine effects on prostate cancer (e.g. saw palmetto and St. John's Wort) 4 weeks prior to randomization.
* Mental incapacity or language barrier precluding adequate understanding or co operation.
* Use of an investigational drug within the last 28 days preceding the Screening Visit or longer if considered to possibly influence the outcome of the current trial.
* Previously participated in any degarelix trial.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Intratumoral androgen levels | Week 12

SECONDARY OUTCOMES:
Prostate tumour morphology related to androgen withdrawal after neo-adjuvant therapy | Week 12

OTHER OUTCOMES:
Serum levels of Androgen Receptor after neo-adjuvant therapy | Baseline, Week 12
Serum level of Follicle Stimulating Hormone (FSH) after neo-adjuvant therapy | Baseline, Week 12
Serum Level of Inhibin-b and GnRH after neo-adjuvant therapy | Baseline, Week 12

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Vancouver General Hospital, Vancouver, British Columbia
  - University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976
- [Derived] Sayyid RK, Evans A, Hersey K, Maloni R, Hurtado-Coll A, Kulkarni G, Finelli A, Zlotta AR, Hamilton R, Gleave M, Fleshner NE. A Phase II, Randomized, Open-Label Study of Neoadjuvant Degarelix versus LHRH Agonist in Prostate Cancer Patients Prior to Radical Prostatectomy. Clin Cancer Res. 2017 Apr 15;23(8):1974-1980. doi: 10.1158/1078-0432.CCR-16-1790. Epub 2016 Oct 18. PMID 27756786